CLINICAL TRIAL: NCT03558672
Title: A Registry to Evaluate the Flexitouch System and Flexitouch Plus for Treatment of Head and Neck Lymphedema
Status: Terminated | Type: Observational
Why Stopped: Low enrollment numbers
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 4060
Record Dates: First submitted 2018-05-10; First posted 2018-06-15 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Lymphedema
Keywords: Flexitouch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Flexitouch system with Head and Neck Garments — Flexitouch system or Flexitouch Plus Head and Neck Treatment, as prescribed

SUMMARY:
The objective of this registry is to evaluate the long term effectiveness of the Flexitouch System and Flexitouch Plus in those with head and neck lymphedema. This outcome data will include information regarding each subject's medical history, symptoms, quality of life, pain, range of motion (ROM), swelling, ease of use, treatment satisfaction, treatment compliance, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A diagnosis of head and/or neck lymphedema
* Must be able and willing to participate in all aspects of the registry and provide informed consent prior to registry participation
* Head and chest measurements within the following:
* Crown of head circumference: ≤ 72 cm
* Chest circumference: ≤ 158 cm
* Prescribed the Flexitouch system or Flexitouch Plus

Exclusion Criteria:

* Uncontrolled hyperthyroidism or parathyroidism (for which endocrinologist recommends against neck compression)
* Carotid sinus hypersensitivity syndrome
* Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke, or amaurosis fugax (monocular visual ischemic symptoms or blindness)
* Symptomatic bradycardia in the absence of a pacemaker
* Internal jugular venous thrombosis (within 3 months)
* Increased intracranial pressure or other contraindications to internal or external jugular venous compression
* Acute radiation dermatitis, unhealed surgical scar, unhealed or open wound(s), or surgical flap less than 6-8 weeks post-operative
* Facial or head and neck dermal metastasis
* Acute facial infection (e.g., facial or parotid gland abscess)
* Any condition in which increased venous and lymphatic return is undesirable
* Heart failure (acute pulmonary edema, decompensated acute heart failure)
* Subject is pregnant or trying to become pregnant
* Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Head and Neck Lymphedema and prescribed the Flexitouch system or Flexitouch Plus system as standard of care treatment
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Iowa ENT Center, West Des Moines, Iowa
  - Charles George VA Medical Center, Asheville, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among therapists and physicians across 4 US sites between September 2018 and March 2020. The first subject was enrolled on September 14, 2018.
Groups:
- Intervention: Participants received either the Flexitouch system or Flexitouch Plus Head and Neck treatment, as prescribed.
Period: Overall Study
Arm/Group | Intervention
Started | 18
Completed | 8
Not Completed | 10
Not completed — Study Early Termination | 10

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes subjects who completed the screening process. This does not include screen failure subjects.
Arm/Group | Intervention
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 62.1 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Race : White or Caucasian | 17
  Race : Black or African American | 1
  Race : Asian | 0
  Race : American Indian or Alaska Native | 2
  Race : Native Hawaiian or Other Pacific Islander | 0
  Race : Other | 0
  Ethnicity: Hispanic or Latino | 1
  Ethnicity: Not Hispanic or Latino | 17

OUTCOME MEASURES:

1. Primary Outcome: Symptom/Problem Improvement From Baseline to 6 Months
Description: To evaluate symptoms based upon the EORTC HN35 questionnaire from baseline to 6 months of treatment with the Flexitouch System or Flexitouch Plus.
  Positive value shows an increase in symptoms/problems. Negative value shows a decrease in symptoms/problems. Percent change is calculated by the difference between scores averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: Although 8 participants had completed the study, only 7 completed all required questionnaires. Therefore, the analysis population only includes the 7 participants who completed the required questionnaires throughout the study.
Measure: Number; unit: percent change in score
Arm/Group | Intervention
Number analyzed (Participants) | 7
percent change in score
  Have you had pain in your mouth? | 14.3
  Have you had pain in your jaw? | 30.0
  Have you had soreness in your mouth? | 17.4
  Have you had a painful throat? | 35.3
  Have you had problems swallowing liquids? | 23.5
  Have you had problems swallowing pureed food? | 53.8
  Have you had problems swallowing solid food? | -7.7
  Have you choked when swallowing? | -20.0
  Have you had problems with your teeth? | 30.0
  Have you had problems opening your mouth wide? | 13.0
  Have you had a dry mouth? | 0.0
  Have you had sticky saliva? | 4.3
  Have you had problems with you sense of smell? | -5.0
  Have you had problems with your sense of taste? | 3.4
  Have you coughed? | -4.2
  Have you been hoarse? | 0.0
  Have you felt ill? | 0.0
  Has your appearance bothered you? | -20.8
  Have you had trouble eating? | 0.0
  Have you had trouble eating in front of family? | 17.6
  Have you had trouble eating in front of people? | -22.2
  Have you had trouble enjoying your meals? | 3.8
  Have you had trouble talking to other people? | -4.8
  Have you had trouble talking on the telephone? | -17.4
  Have you had trouble social contact with family? | -29.4
  Have you had trouble social contact with friends? | -19.0
  Have you had trouble going out in public? | -23.8
  Have you had trouble having physical contact? | -35.3
  Have you felt less interest in sex? | 0.0
  Have you felt less sexual enjoyment? | -14.8
  Have you used pain killers? | 28.6
  Have you taken any nutritional supplements? | 50.0
  Have you used a feeding tube? | -50.0
  Have you lost weight? | -20.0
  Have you gained weight? | 57.1

2. Primary Outcome: Function (Range of Motion) Improvement From Baseline to 6 Months
Description: To evaluate function based upon cervical and shoulder range of motions measurements from baseline to 6 months of treatment with the Flexitouch System or Flexitouch Plus.
  Positive value shows an increase in Function/Range of Motion. Negative value shows a decrease in Function/Range of Motion. Percent change is calculated by the difference between measurements averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: Analysis includes the 8 participants who completed the study required visits and assessments.
Measure: Number; unit: percent change in measurement
Arm/Group | Intervention
Number analyzed (Participants) | 8
percent change in measurement
  Cervical: Flexion | 3.7
  Cervical: Extension | 28.9
  Cervical: Right Lateral | 1.5
  Cervical: Left Lateral | 15.9
  Cervical: Right Rotation | 28.5
  Cervical: Left Rotation | 7.8
  Shoulder: Right Flexion | -2.0
  Shoulder: Right Abduction | 12.6
  Shoulder: Left Flexion | -1.9
  Shoulder: Left Abduction | 2.6
  Mouth: Open | 0.6

3. Secondary Outcome: Changes in Health-related Quality of Life From Baseline to 6 Months
Description: Subject Quality of Life will be assessed using EORTC C30 questionnaire. Positive value shows an decrease in quality of life. Negative value shows a increase in quality of life. Percent change is calculated by the difference between scores averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: as for outcome 1
Measure: Number; unit: percent change in score
Arm/Group | Intervention
Number analyzed (Participants) | 7
percent change in score
  Do you have trouble doing strenuous activities? | -17.2
  Do you have any trouble taking a long walk? | 0.0
  Do you have trouble taking a short walk? | -12.5
  Do you need to stay in bed or a chair during day? | 0.0
  Do you need help eating, dressing, washing? | 40.0
  Were you limited in work or other day activities? | 4.3
  Were you limited in hobbies or leisure activities? | 8.3
  Were you short of breath? | 6.3
  Have you had pain? | 0.0
  Did you need to rest? | 21.1
  Have you had trouble sleeping? | -12.5
  Have you felt weak? | 0.0
  Have you lacked appetite? | 5.0
  Have you felt nauseated? | 10.0
  Have you vomited? | 0.0
  Have you been constipated? | -18.8
  Have you had diarrhea? | 7.1
  Were you tired? | 0.0
  Did pain interfere with daily activities? | 0.0
  Have you had difficulty concentrating? | -5.9
  Did you feel tense? | 0.0
  Did you worry? | 10.5
  Did you feel Irritable? | 0.0
  Did you feel depressed? | 25.0
  Have you had difficulty remembering things? | 0.0
  Has condition/treatment interfered with family? | -18.2
  Has condition/treatment interfered socially? | 0.0
  Has condition/treatment caused difficult finances? | -4.8

4. Secondary Outcome: Changes in Health-related Quality of Life-Overall From Baseline to 6 Months
Description: Subject overall health and quality of life in the past week-EORTC C30. Positive value shows an increase in quality of life/overall health. Negative value shows a decrease in quality of life/overall health. Percent change is calculated by the difference between scores averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: as for outcome 1
Measure: Number; unit: % change from baseline to 6 months
Arm/Group | Intervention
Number analyzed (Participants) | 7
% change from baseline to 6 months
  Overall health during the past week | 4.3
  Overall quality of life during the past week | 0.0

5. Secondary Outcome: Changes in Pain From Baseline to 6 Months
Description: Pain will be assessed using the VAS Pain Scale. Positive value shows an increase in pain. Negative value shows a decrease in pain. Percent change is calculated by the difference between scores averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: as for outcome 1
Measure: Number; unit: percent change in score
Arm/Group | Intervention
Number analyzed (Participants) | 7
percent change in score | 47.5

6. Secondary Outcome: Change in Swelling From Baseline to 6 Months
Description: Swelling will be assessed using the ALOHA measurement protocol. Positive value shows an increase in swelling. Negative value shows a decrease in swelling. Percent change is calculated by the difference between swelling measurements averaged at 6 months versus baseline.
Time Frame: Percent Changes between Baseline and 6 months will be assessed
Population: Analysis includes the 8 participants who completed the study required visits and assessments.
Measure: Number; unit: percent change in swelling measurements
Arm/Group | Intervention
Number analyzed (Participants) | 8
percent change in swelling measurements
  Lower Neck Circumference | -3.0
  Upper Neck Circumference | -2.1
  Ear to Ear Length | -2.6

7. Secondary Outcome: Ease of Use/Satisfaction
Description: Both Ease of Use/Satisfaction will be assessed by survey. Percentage of each response captured.
Time Frame: Assessed at 6 months
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Intervention
Number analyzed (Participants) | 7
percent of participants
  Very difficult to use Flexitouch garments | 0.0
  Difficult to use Flexitouch garments | 0.0
  Neither easy nor difficult with Flexitouch garment | 14.3
  Easy to use Flexitouch garments | 57.1
  Very easy to use Flexitouch garments | 28.6
  Very difficult to use Flexitouch controller | 0.0
  Difficult to use Flexitouch controller | 0.0
  Neither easy nor difficult-Flexitouch controller | 0.0
  Easy to use Flexitouch controller | 42.9
  Very easy to use Flexitouch controller | 57.1
  Very uncomfortable treatment by Flexitouch system | 0.0
  Uncomfortable treatment by Flexitouch system | 0.0
  Neither uncomfortable nor comfortable treatment | 0.0
  Comfortable treatment by Flexitouch system | 57.1
  Very comfortable treatment by Flexitouch system | 42.9
  Very dissatisfied overall with Flexitouch system | 0.0
  Dissatisfied overall with Flexitouch system | 0.0
  Neither dissatisfied nor satisfied overall | 0.0
  Satisfied overall with Flexitouch system | 28.6
  Very satisfied overall with Flexitouch system | 71.4
  Yes, would recommend Flexitouch system to others | 100
  No,would not recommend Flexitouch system to others | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on participants who received and were trained on the device from the 2 week visit until 6 month visit or study exit.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=18)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Lingual villosa (Skin and subcutaneous tissue disorders) | 1 (1)
Osteomylelitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated in regards to slow enrollment; there were no safety issues presented. The variability in the small N (N=8) provide inconclusive evidence and non analyzable outcome measure from this incomplete data cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03558672/Prot_SAP_000.pdf